CLINICAL TRIAL: NCT02125812
Title: Adjunctive Systemic Administration of Moxifloxacin in the Treatment of Aggressive Periodontitis: Double-blind Controlled Clinical Trial
Brief Title: Adjunctive Systemic Administration of Moxifloxacin in the Treatment of Aggressive Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Facultad Nacional de Salud Publica (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Carlos Martin Ardila Medina, Titular Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Aggressive Periodontitis
Keywords: Aggressive Periodontitis; antimicrobial(s); microbiology
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- scaling and root planing (Placebo Comparator): scaling and root planing
  Interventions: Other: scaling and root planing
- scaling and systemic moxifloxacin (Experimental): scaling and root planing combined with systemic moxifloxacin
  Interventions: Other: scaling and systemic moxifloxacin

INTERVENTIONS:
Other: scaling and systemic moxifloxacin — scaling and root planing (SRP) combined with systemic moxifloxacin
  Arms: scaling and systemic moxifloxacin
Other: scaling and root planing — scaling and root planing
  Arms: scaling and root planing

SUMMARY:
The adjunctive use of systemically administered antibiotics has been shown to provide a better clinical outcome, particularly in terms of probing depth (PD) reduction and attachment-level gain than SRP in subjects with Aggressive Periodontitis.

The overall objective of this study is to evaluate the clinical and microbiological efficacy of moxifloxacin as an adjunct to scaling and root planing versus scaling and root planing over placebo in the treatment of aggressive periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* under 30 years old and systemically healthy, with at least 20 teeth present. Be willing to participate in the study which is corroborated by signing the informed consent form.

Commit to attend post-therapeutic controls and stop drinking alcohol during the time of ingestion of antibiotics.

Exclusion Criteria:

* Subjects in whom are contraindicated or with hypersensitivity to quinolones - Subjects who have undergone periodontal, surgical or mechanical antibiotic therapy six months before the start of the study according to interrogation.

Women in pregnancy or lactation, corroborated with previous medical history and medical consultation.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
probing depth | six months

SECONDARY OUTCOMES:
clinical attachment level and probing depth | 6 moths

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Ardila, Ph.D, Principal Investigator — Universidad de Antioquia
Locations (1):
- Faculty of Dentistry, Departamento de Antioquia, Medellin, Colombia

REFERENCES:
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- See also: Universidad de Antioquia — http://odontologia.udea.edu.co